CLINICAL TRIAL: NCT00603135
Title: Intravenous Levetiracetam as First-line Anticonvulsive Treatment in Patients With Non-convulsive Status Epilepticus
Acronym: Keppra
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Hospital, Basel, Switzerland, Dr. med. Stephan Rüegg, Neurology (Other); Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Dr. med. Stephan Rüegg, Neurology,University Hospital Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNeuro_Keppra_; EKBB 272/27
Record Dates: First submitted 2007-11-13; First posted 2008-01-28 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Status Epilepticus, Non-Convulsive
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: first-line i/v-levetiracetam

INTERVENTIONS:
Drug: first-line i/v-levetiracetam — No effect after 30 min, standard therapy with f.e. lorazepam for NCSE

SUMMARY:
Status epilepticus (SE) represents the most common life-threatening neurological emergency requiring treatment on an intensive care unit. The incidence in Western European countries is about 12-18/100'000. Immediate and effective treatment of SE is obviously essential because of the deleterious effects of continuous seizures on the brain and the whole organism. Guidelines emphasize the use of benzodiazepines (BZD) as first-line anticonvulsive drugs. Alternatively, i/v Phenytoin (PHE), fosphenytoin (FOS), and valproate (VPA) were also tested as first-line anticonvulsants in SE. Direct comparison of PHE with lorazepam (LZP) showed significant superiority of LZP (evidence class I). Other trials i/v PHE or -VPA are of evidence class III or IV. BZD, VPA, and PHE have clinical and pharmacological disadvantages. BZD may cause respiratory depression or sedation and may be not suitable for patients with COPD or ambiguous in patients with BZD addiction. Some compounds also may induce tachyphylaxis or accumulate under concomitant renal failure. PHE has saturable metabolism subject to Michaelis-Menten kinetics increasing the risk of overdosing in an acute setting causing liver damage, serious cardiac arrhythmias, hypotension, cerebellar degeneration, peripheral neuropathy and local/systemic skin reactions. Although of unequivocal efficacy, PHE should no longer be used for long-term because of its adverse effects after chronic administration (irreversible cerebellar degeneration causing debilitating ataxia, painful polyneuropathy, and osteopenia increasing the risk of fractures). Metabolism by and self-induction of the hepatic CYP450 system make PHE prone to interactions with several other drugs, notably other antiepileptics. VPA may cause liver failure, hemorrhagic complications, pancreatitis, and hyperammonemic encephalopathy. To summarize, these three first-line agents for the treatment of SE may cause serious side effects in several patients with SE.

Levetiracetam (LEV) is broad-spectrum antiepileptic drug. It binds to the presynaptic vesicular protein 2A abundantly present in different regions of the brain; LEV presynaptically modulates transmitter release, but the exact mechanism(s) remain unclear. Data also revealed that LEV stabilizes GABAA receptors upon repetitive activation what is important in treatment of SE because GABAA receptors undergo significant changes of subunit conformation within minutes after sustained activation like during SE. These changes render GABAA receptors the less anticonvulsive, the longer SE lasts. Levetiracetam has a favorable pharmacological profile with large safety margins. Its partly extrahepatic hydrolyzation bypasses the CYP450 system; renal excretion is 60-70% unchanged, and 23-27% metabolized. Dosage needs adjustment when renal function is impaired. LEV lacks interactions with any drugs yet. Drowsiness is the most common side-effect while respiration, liver and kidney function, and the blood system are not affected. LEV shows an important clinical effect even after the first dose and maximal efficacy within the first week of drug-intake. The favorable clinico-pharmacological profile predilects LEV for the first-line treatment of SE, especially in patients with multi-organ failure, sepsis, coma etc.. About 10 % of comatous patients may be in non-convulsive SE (NCSE) on ICU's. These patients are under polymedication whereby interactions of the anticonvulsants approved yet for the treatment of NCSE with their other drugs may have fatal effects. Conversely, non-interacting anticonvulsants would represent an advantage for the treatment of NCSE for these patients.

Recently, the i/v formulation of LEV was approved by the FDA for the use in patients, but not specifically for the treatment of SE. Data about the single-dose bioavailability of i/v-LEV in comparison to oral tablets as well as multiple-dose pharmacokinetics and tolerability in healthy subjects were recently published. In addition, the administration of i/v-LEV dosages ranging from 2000-4000 mg within 15 minutes and of dosages ranging from 1500-2500 mg within 5 minutes was safe and well tolerated, and led to efficacious drug levels in a randomized, single-blind, placebo-controlled safety and pharmacokinetic study in healthy volunteers.

Slight somnolence is expected to be the only adverse effect of i/v LEV, sharply contrasting with the sedation up to coma after i/v benzodiazepines. Thus, even severely ill patients will be accessible to neurological tests under LEV which is a big advantage in this clinical difficult setting of NCSE.

I-v LEV is considered an ideal candidate for the first-line use (before benzodiazepines) in patients with NCSE, especially in those with important comorbidity and concomitant polymedication. Thus, we would like to test the feasibility, safety, and efficacy of i/v-LEV as first-line medication in a open-label, single-center, prospective pilot study as outlined below.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older with NCSE. NCSE includes the following subtypes:

  * simple partial NCSE
  * complex partial status epilpeticus
* Absence status
* NCSE in critical illness
* Written informed consent should be signed.

Exclusion Criteria:

* Age below 20
* Known intolerance to the study drug levetiracetam
* Known pregnancy
* Postanoxic SE
* Subtle SE

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy/ Clinical and/or electroencephalographic cessation of SE | 30 min

SECONDARY OUTCOMES:
safety | 48 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Rüegg, MD, Principal Investigator — Neurology; Stephan Rüegg, MD, Study Chair — Neurology
Locations (1):
- University Hospital Basel, Basel, Basel, Switzerland

REFERENCES:
- [Background] Rupprecht S, Franke K, Fitzek S, Witte OW, Hagemann G. Levetiracetam as a treatment option in non-convulsive status epilepticus. Epilepsy Res. 2007 Mar;73(3):238-44. doi: 10.1016/j.eplepsyres.2006.10.011. Epub 2006 Dec 8. PMID 17161587
- [Result] Ruegg SJ, Dichter MA. Diagnosis and Treatment of Nonconvulsive Status Epilepticus in an Intensive Care Unit Setting. Curr Treat Options Neurol. 2003 Mar;5(2):93-110. doi: 10.1007/s11940-003-0001-4. PMID 12628059
- [Result] Ramael S, Daoust A, Otoul C, Toublanc N, Troenaru M, Lu ZS, Stockis A. Levetiracetam intravenous infusion: a randomized, placebo-controlled safety and pharmacokinetic study. Epilepsia. 2006 Jul;47(7):1128-35. doi: 10.1111/j.1528-1167.2006.00586.x. PMID 16886975
- [Result] Ramael S, De Smedt F, Toublanc N, Otoul C, Boulanger P, Riethuisen JM, Stockis A. Single-dose bioavailability of levetiracetam intravenous infusion relative to oral tablets and multiple-dose pharmacokinetics and tolerability of levetiracetam intravenous infusion compared with placebo in healthy subjects. Clin Ther. 2006 May;28(5):734-44. doi: 10.1016/j.clinthera.2006.05.004. PMID 16861095